CLINICAL TRIAL: NCT07308340
Title: Clinical Study on Rapid Identification of Infectious Pathogens in Severe Pneumonia Patients Based on Bronchoscopic Imaging and Lung CT Guidance
Brief Title: Rapid Identification of Infectious Pathogens in Severe Pneumonia Guided by Bronchoscopic Imaging and Lung CT
Acronym: IMG-GUIDE-IP
Status: Not yet recruiting | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Hongxiang Li, Chief Physician, Associate Professor, PhD, The First Hospital of Jilin University
Other Study IDs: IPID-2026
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-12

CONDITIONS: Severe Pneumonia
Keywords: Severe Pneumonia; Infectious Pathogen Identification; Bronchoscopic Imaging; Lung CT; Retrospective Cohort Study
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe Pneumonia Patients with Dual Diagnostic Assessments: This retrospective cohort includes patients diagnosed with severe pneumonia who were admitted to the study institution between 2024 and 2025 (recruitment will be extended 6-12 months if fewer than 400 patients are enrolled). All patients in this cohort underwent two diagnostic procedures (standalone lung CT, and bronchoscopic imaging combined with lung CT) during their clinical management. The cohort is designed for self-controlled comparison: diagnostic accuracy of the two methods for infectious pathogen identification will be analyzed to verify the value of the combined imaging approach.
  Interventions: Diagnostic Test: Standalone Lung CT for Severe Pneumonia Diagnosis; Diagnostic Test: Bronchoscopic Imaging + Lung CT for Severe Pneumonia diagnosis

INTERVENTIONS:
Diagnostic Test: Standalone Lung CT for Severe Pneumonia Diagnosis — Standard chest CT scan (including plain scan and/or enhanced scan as clinically needed) performed to evaluate pulmonary lesion location, scope, and imaging features (e.g., consolidation, ground-glass opacity). The CT findings will be used to preliminarily infer the presence of infectious pathogens and guide initial clinical judgment.
Diagnostic Test: Bronchoscopic Imaging + Lung CT for Severe Pneumonia diagnosis — Based on pre-existing lung CT images (to locate lesions), flexible bronchoscopy is performed to directly observe mucosal changes in the tracheobronchial tree (e.g., congestion, edema, exudation). Bronchoscopic imaging features are combined with CT findings to comprehensively judge the type of infectious pathogen (e.g., bacterial vs. viral) and improve diagnostic accuracy.

SUMMARY:
Severe pneumonia requires rapid and accurate diagnosis for targeted treatment, but single lung CT has limitations in identifying pathogens and distinguishing infectious/non-infectious etiologies. This is a retrospective self-controlled study enrolling patients diagnosed with severe pneumonia at the institution between 2024 and 2025 (recruitment will be extended 6-12 months if fewer than 400 patients are enrolled), all of whom underwent both single lung CT and bronchoscopy-combined CT examinations.

Clinical data will be collected retrospectively, including demographic information, bronchoscopic mucosal findings (e.g., congestion, exudation), lung CT lesion characteristics (e.g., consolidation, ground-glass opacity), and gold standard diagnostic results (pathogenic detection or clinical comprehensive diagnosis). The core objective is to compare the diagnostic precision between single lung CT and bronchoscopy-combined CT, focusing on accuracy, sensitivity, and specificity across three etiological subtypes (bacterial/fungal, viral, non-infectious).

Bronchoscopy complements CT by directly visualizing airway mucosal changes, while CT provides panoramic views of pulmonary lesions. Their combination is hypothesized to improve diagnostic accuracy. The findings aim to optimize diagnostic strategies for severe pneumonia, guiding clinicians to select more effective imaging approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the study institution between January 2024 and December 2025, with a clinical diagnosis of severe pneumonia (consistent with the diagnostic criteria of the Chinese Guidelines for the Diagnosis and Treatment of Community-Acquired Pneumonia.
* Patients who underwent both standalone lung CT examination and bronchoscopic imaging examination during hospitalization; complete imaging reports and bronchoscopy operation records are available.
* Patients who completed at least one type of microbial standard test (as defined in Primary Outcome Measure: e.g., pathogen culture, nucleic acid detection, GM test); complete test reports are available.
* Medical Records: Complete electronic medical records are available, including demographic information (age, gender), clinical symptoms, treatment regimens, and prognosis data (length of hospital stay, in-hospital mortality).

Exclusion Criteria:

* Imaging/Microbial Data Deficiency: Patients with incomplete imaging data (e.g., missing lung CT images, unrecorded bronchoscopic mucosal changes) or unavailable microbial gold standard test results.
* Bronchoscopy Contraindications: Patients who underwent bronchoscopic imaging for non-diagnostic purposes (e.g., foreign body removal, hemostasis) or had bronchoscopy-related complications (e.g., severe hemorrhage, pneumothorax) that affected examination completion.
* Duplicate Enrollment: Patients who were admitted multiple times for severe pneumonia during the study period; only the first admission is included to avoid duplicate data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients (≥18 years old) admitted to the study institution between January 2024 and December 2025, with a confirmed diagnosis of severe pneumonia (per Chinese clinical guidelines for community-acquired or hospital-acquired pneumonia). All included patients must have undergone both standalone lung CT and bronchoscopic imaging (CT-guided) during hospitalization, with complete imaging records. They also need to have completed at least one microbial gold standard test (e.g., pathogen culture, nucleic acid detection) with available reports, and intact electronic medical records (demographics, treatment, prognosis).
  Patients are excluded if they have incomplete imaging/microbial data, bronchoscopy for non-diagnostic purposes, duplicate admissions, or are under 18 years old.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Two Imaging Methods for Infectious Pathogens in Severe Pneumonia | Data collection will be completed retrospectively within 6 months after the last patient (admitted by 2025) is included; diagnostic accuracy analysis will be finished within 6 months after data collection.
  For each patient in the cohort, the diagnostic results of standalone lung CT and bronchoscopic imaging + lung CT will be compared with the "standard for pathogen diagnosis" (e.g., pathogen culture, nucleic acid detection, serological testing) to calculate two key indicators: 1. Sensitivity: The proportion of patients with positive gold standard results that are correctly identified as positive by the diagnostic method; >2. Specificity: The proportion of patients with negative gold standard results that are correctly identified as negative by the diagnostic method. primary goal is to verify whether the combined imaging method (bronchoscopy + CT) has higher sensitivity and specificity than standalone CT for identifying infectious pathogens (including bacteria, fungi, and viruses).

IPD SHARING:
Plan to Share IPD: Yes
We plan to share de-identified individual participant data (IPD) that includes:
  Demographic information (e.g., age, gender); Baseline clinical characteristics (e.g., disease stage, results of relevant laboratory tests); Intervention-associated data (e.g., diagnostic findings from computed tomography (CT) alone and combined with bronchoscopy); Outcome measures (the accuracy of diagnosis for severe pneumonia); Safety data (e.g., documentation of adverse events). To safeguard participant privacy, all shared data will be fully de-identified by removing direct identifiers (e.g., full name, contact details, medical record number).
Supporting Information: Study Protocol, SAP, CSR